CLINICAL TRIAL: NCT03548623
Title: Patient Preference in Blood Pressure Therapy: Questioning of Patients With Hypertension
Brief Title: Patient Preference in Blood Pressure Therapy
Status: Completed | Type: Observational
Sponsor: Roland E. Schmieder (Other)
Collaborators: Institute for Preventive Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Roland E. Schmieder, Full Professor of Medicine, University of Erlangen-Nürnberg Medical School
Organization: University of Erlangen-Nürnberg Medical School (Other)
Other Study IDs: CRC2017PPiB
Record Dates: First submitted 2018-04-23; First posted 2018-06-07 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Arterial Hypertension
Keywords: Hypertension; renal denervation; preference; shared decision making
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Written surveys of patients with high blood pressure are designed to determine how they would likely decide if, in addition to taking medication, they had another option to treat their hypertension.

The alternative treatment option is renal sympathetic denervation using catheter ablation. This new treatment method is not yet used in the standard care. Currently, studies are being conducted in specific centers to demonstrate the efficacy of this treatment.

Questionnaires are used to determine the preference of patients for one or the other option of hypertension treatment. So far, there are no findings.

ELIGIBILITY:
Inclusion Criteria:

* untreated Hypertension
* treated Hypertension with one or more medications

Exclusion Criteria:

* illiteracy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * male and female
  * > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Preference of treatment | 3 months
  Questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Preventive Medicine, Nuremberg, Germany

IPD SHARING:
Plan to Share IPD: No